CLINICAL TRIAL: NCT04079582
Title: Outcomes of a Higher vs. Lower Hemodialysate Magnesium Concentration: A Pragmatic Cluster-randomized Clinical Trial in Hemodialysis Centres
Brief Title: Outcomes of a Higher vs. Lower Hemodialysate Magnesium Concentration (Dial-Mag Canada)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: ICES (Industry); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R-13-999
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Kidney Diseases; End-Stage Kidney Disease; Hemodialysis
Keywords: Dialysate Magnesium; Kidney Disease; Renal Insufficiency, Chronic; Kidney Failure, Chronic; Cluster Randomized Controlled Trial
MeSH Terms: conditions — Kidney Diseases; Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Higher dialysate magnesium (Experimental)
  Interventions: Other: Dialysate magnesium formulation of 1.5 mEq/L (0.75 mmol/L).
- Lower dialysate magnesium (Active Comparator)
  Interventions: Other: Dialysate magnesium formulation of ≤1.0 mEq/L (≤0.5 mmol/L).

INTERVENTIONS:
Other: Dialysate magnesium formulation of 1.5 mEq/L (0.75 mmol/L). — (Dialysate magnesium concentration currently used in Canada and the United States)
  Arms: Higher dialysate magnesium
Other: Dialysate magnesium formulation of ≤1.0 mEq/L (≤0.5 mmol/L). — (Dialysate magnesium concentration currently used in Canada and the United States)
  Arms: Lower dialysate magnesium

SUMMARY:
Many patients on hemodialysis have low levels of magnesium. Magnesium is needed to keep the heart, kidneys, and other organs working properly. Patients with low serum magnesium concentration have a higher risk of death, heart issues, muscle cramps and fractures. There are several reasons why patients on dialysis have low levels of magnesium-these include poor diet, medication interference, and the dialysis procedure itself, which leaches small amounts of magnesium from the blood during each treatment.

One way to make sure that patients on dialysis are getting enough magnesium is to increase its concentration in the dialysate. The investigator would like to do a randomized controlled trial to determine the effect of increasing the concentration of magnesium in the dialysate on the risk of people on dialysis dying or being admitted to the hospital due to heart issues. The investigator thinks increasing the magnesium in the dialysate will help patients live longer, have fewer hospitalisations related to heart disease and patients may also experience less cramping associated with dialysis.

This simple adjustment to the dialysis procedure can be done at little cost and may even reduce overall healthcare costs. If the investigator can show that increasing magnesium in the dialysate improves patients' health, then it could become the standard of care for all patients on dialysis.

DETAILED DESCRIPTION:
1. Statement of the health problem or issue

   In end-stage kidney disease, dialysis is needed to remove toxins and electrolytes that would otherwise accumulate in a patient's blood. The fluid used in dialysis, the dialysate, contains magnesium, and the lower the concentration of dialysate magnesium, the more magnesium is removed from a patient's body during dialysis. Understanding the optimal amount of magnesium to include in the dialysate is crucial as magnesium regulates more than 300 enzymes in the body and is vital to heart, muscle, and bone health.

   In Canada, the dialysate is prepared by central suppliers and contains magnesium in concentrations of 0.38, 0.5, or 0.75 mmol/L. In the absence of clinical trial evidence, there is no consensus on what magnesium concentration is best, and all 3 concentrations are used today in Canadian hemodialysis centres.
2. Objective of the project

   In outpatients receiving conventional hemodialysis, to determine if providing a higher versus lower dialysate magnesium concentration (0.75 vs. ≤0.5 mmol/L) as a centre policy alters outcomes important to patients and their providers.
3. Outline

   This is a pragmatic, two-arm, parallel-group, cluster-randomized, open-label, multicentre, comparative-effectiveness trial embedded into routine care in hemodialysis centres in Canada. Centres have been randomized to, and are receiving a dialysate magnesium concentration of 0.75 mmol/L or ≤0.5 mmol/L in the intervention and control groups, respectively. Patients receiving maintenance hemodialysis at these centres will be followed for study outcomes during the trial follow-up period.

   The trial is highly pragmatic to facilitate high intervention adherence and extensive uptake of the findings; pragmatic features include (i) broad eligibility criteria and a large representative sample of hemodialysis centres and patients, (ii) intervention implementation within routine clinical care delivered by dialysis unit personnel rather than researchers, (iii) follow-up of patient outcomes using routinely collected data sources, (iv) an intent-to-treat analysis using all available data, and (v) outcomes highly relevant to patients.
4. What is unique/innovative about the project?

   The investigator usually needs to study a large number of patients in a clinical trial to reliably understand the effects of a treatment. Normally, a study with 15,000 patients would cost more than $15 million dollars to conduct; however, this study will provide a reliable answer to the question being asked and cost less than $4 million. This is because the majority of data is already being collected by the healthcare system. For example, when a patient is hospitalized for a heart attack or stroke, this information is recorded in a secure healthcare database. The investigator will be able to analyze these healthcare data at the end of the study (and link patient outcomes to the type of dialysis treatment received (i.e. treatment or control). This innovative study design means that the study will be much larger (but cost much less) than a traditional clinical trial.

   This pragmatic trial includes all patients who receive chronic in-centre hemodialysis patients in participating centres. High-risk patients with multiple comorbidities, including cognitive impairments or disabilities, who are often excluded from trials because of their high-risk status are eligible for participation in the Dialysate Magnesium trial. By including patients from a variety of medical, ethnic, geographic, and socioeconomic backgrounds, the results of the trial should be broadly generalizable.
5. What is the impact of the proposed research?

For patients with severe kidney failure (10,000 in Ontario and >2 million worldwide), hemodialysis provides a life-saving treatment option; however a tragic 20-40% of patients die within one year of starting hemodialysis. The dialysate is a critical component of hemodialysis, yet little evidence is available to guide its optimal formulation. Dialysate magnesium in particular has received little scientific attention until recently, with new research suggesting that a higher dialysate magnesium concentration may benefit patients. Outcomes that may be improved include mortality, cardiovascular outcomes, and muscle cramps.

While it is possible to raise the concentration of serum magnesium through oral supplements, using dialysis to do this is simpler and safer. It has no additional cost, does not add to a patient's pill burden, is not dependent on an adherent patient taking their pills, and avoids the gastrointestinal side effects of oral magnesium supplements.

If the investigator is able to demonstrate that a higher dialysate magnesium concentration improves patient outcomes, this formulation can be readily adopted to improve the care of ∼2 million patients receiving hemodialysis worldwide.

ELIGIBILITY:
Inclusion Criteria: This pragmatic cluster randomized controlled trial has only two inclusion criteria:

1. The hemodialysis centre, or a group of hemodialysis centers combined into one cluster, must care for at least 15 outpatients being treated with in-centre maintenance hemodialysis.
2. The medical director of the hemodialysis centre must be willing for their centre to be randomized and to adopt the allocated dialysate Mg protocol as their standard solution for the duration of the trial.

Exclusion Criteria:

* The centre, or group of hemodialysis centres cares for less than 15 patients being treated with conventional in-centre hemodialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25000 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of cardiovascular-related hospitalization and all-cause mortality | Three to Four Years
  Cardiovascular-related hospitalization (for myocardial infarction, ischemic stroke, or congestive heart failure) will be ascertained using primary discharge ICD-10 diagnosis codes in the Canadian Institute for Health Information's Discharge Abstract Database. All-cause mortality is recorded with over 99% accuracy in our data sources.

SECONDARY OUTCOMES:
Key secondary outcome - patient-reported muscle cramps | Three to Four Years
  Patients will be able to voluntarily and anonymously answer a question on muscle cramps to describe on average how much this symptom bothered them in the past week. Responses will be recorded on a 10-point scale, with 0 indicating absence of the symptom and 10 indicating the symptom is at its worst. The question will be made available in the dialysis centre approximately twice a year. No patient identifiers will be collected and this outcome will be assessed at the level of the centre.
Components of the primary composite outcome | Three to Four Years
  Each component of the primary composite outcome (all-cause mortality and hospitalizations for myocardial infarction, ischemic stroke, and congestive heart failure) will be examined separately.

CONTACTS AND LOCATIONS:
Overall Officials: Amit X Garg, PhD, MD, Principal Investigator — ICES, Lawson, London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dial-Mag Investigator Writing Committee*; Killin L, Bohm C, Harris C, MacRae JM, Shah N, Thompson S, Tonelli M, Luo B, Sontrop JM, Acedillo RR, Al-Jaishi AA, Anderson S, Antonsen J, Bagga A, Beaubien E, Berry D, Blake PG, Brown PA, Bueti J, Chan CT, Cote B, Cowan AC, Cuerden MS, Day NE, Dev V, Dhruve M, Djurdjev O, Gregor L, Hiremath S, Joseph G, Kammila S, Kiaii M, Kumar Kolusu E, Lacson E Jr, Mazurat A, Molnar AO, Nathoo B, Nistico A, Oliver MJ, Pandeya S, Parmar MS, Perkins D, Quinn K, Romann A, Sasal J, Shulman T, Silver SA, Singh A, Louis IS, Steele A, Tangri N, Ting RH, Vorster H, Wadehra DB, Wald R, Walters J, Whitlock RH, Yao S, Zacharias J, Garg AX. Outcomes of Adopting a Higher Versus Lower Concentration of Hemodialysate Magnesium as a Center-Wide Policy (Dial-Mag): A Clinical Research Protocol of a Pragmatic, Registry-Based, Cluster Randomized Trial. Can J Kidney Health Dis. 2025 Dec 9;12:20543581251385011. doi: 10.1177/20543581251385011. eCollection 2025. PMID 41393273